CLINICAL TRIAL: NCT02123628
Title: Six- Versus Twelve-Week Therapy for Non-Surgically-Treated Diabetic Foot Osteomyelitis: A Multicenter Open-Label Controlled Randomized Study
Brief Title: Antibiotic Treatment Duration for Non-Surgically-Treated Diabetic Foot Osteomyelitis
Acronym: C H R O N O S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-00625-14
Record Dates: First submitted 2014-04-15; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus
Keywords: diabetic foot osteomyelitis, antibiotic treatment duration
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rifampin; Levofloxacin; Doxycycline; Trimethoprim, Sulfamethoxazole Drug Combination; Fusidic Acid; Linezolid; Ciprofloxacin; Cefotaxime; Ceftriaxone; Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- antibiotic therapy (Active Comparator): patients are treated with a 6 week-duration of antibiotic therapy :
  * Rifampin IP and PO twice daily, 10mg/kg /12H
  * Levofloxacin IV and PO 500-750mg once daily
  * Doxycycline PO 200mg once daily
  * Trimethoprim- sulfamethoxazole IV and PO 800/160mg thrice daily
  * Fusidic acid PO 500mg twice daily
  * Linezolid IV and PO 600mg twice daily
  * Ciprofloxacin IV and PO 750to 1000mg/12h
  * Cefotaxime IV 100mg/kg in three IV infusions daily
  * Ceftriaxone IV,intramuscularly or subcutaneously 2g once daily
  * Cefepime IV ou intra-muscularly 2g /8-12h
  Interventions: Drug: duration of the antibiotic therapy
- 12 week-duration of antibiotic therapy (Active Comparator): patients are treated with a 12 week-duration of antibiotic therapy :
  * Rifampin IP and PO twice daily, 10mg/kg /12H
  * Levofloxacin IV and PO 500-750mg once daily
  * Doxycycline PO 200mg once daily
  * Trimethoprim- sulfamethoxazole IV and PO 800/160mg thrice daily
  * Fusidic acid PO 500mg twice daily
  * Linezolid IV and PO 600mg twice daily
  * Ciprofloxacin IV and PO 750to 1000mg/12h
  * Cefotaxime IV 100mg/kg in three IV infusions daily
  * Ceftriaxone IV,intramuscularly or subcutaneously 2g once daily
  * Cefepime IV ou intra-muscularly 2g /8-12h
  Interventions: Drug: duration of the antibiotic therapy

INTERVENTIONS:
Drug: duration of the antibiotic therapy
  Other Names: - Rifampin; - Levofloxacin; - Doxycycline; - Trimethoprim- sulfamethoxazole; - Fusidic acid; - Linezolid; - Ciprofloxacin; - Cefotaxime; - Ceftriaxone; - Cefepime

SUMMARY:
The purpose of the study is to compare the efficacy and tolerance of 6- versus 12-week antibiotic therapy in patients with diabetic foot osteomyelitis treated medically.

DETAILED DESCRIPTION:
The aim of this randomized multicenter clinical study is to compare the efficacy and tolerance of 6 versus 12-week antibiotic treatment in patients with diabetic foot osteomyelitis treated medically as no equivalent data are currenty available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients treated non-surgically (i.e. without amputation or resection of the infected bone) for an osteomyelitis of the foot complicating a neuropathic foot without ischemia of the foot defined as the absence of any pedal pulse. Patients aged of 18 years or more were included if they had type 2 diabetes and osteomyelitis of the foot (i.e.below the ankle).

Exclusion Criteria:

* Patients with gangrene or who require bone resection or amputation when osteomyelitis of the foot was diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was the proportion of patients of each group with remission of diabetic foot osteomyelitis at the end of follow-up. | one year
  Remission was defined as the absence of any sign of infection at the initial or a contiguous site, evaluated at least one year after the end of antibiotic treatment (ie at the end of follow-up), with neither a new infectious episode nor the need for orthopedic surgery of the foot at either of these sites during the treatment and follow-up period.

SECONDARY OUTCOMES:
tolerance to treatment in each group of patients | 6 or 12 weeks
  number of episodes of adverse events attributable to the antibiotic treatment recorded in each group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Senneville, MD, PhD, Study Director — Dron Hospital of Tourcoing France; Alina Tone, MD, Principal Investigator — Dron Hospital Tourcoing France
Locations (1):
- Dron Hospital, Tourcoing, Nord, France

REFERENCES:
- [Derived] Tone A, Nguyen S, Devemy F, Topolinski H, Valette M, Cazaubiel M, Fayard A, Beltrand E, Lemaire C, Senneville E. Six-week versus twelve-week antibiotic therapy for nonsurgically treated diabetic foot osteomyelitis: a multicenter open-label controlled randomized study. Diabetes Care. 2015 Feb;38(2):302-7. doi: 10.2337/dc14-1514. Epub 2014 Nov 20. PMID 25414157